CLINICAL TRIAL: NCT07225257
Title: RETURN: Recovery of Physical Function After Critical Illness In Older Adults
Brief Title: Recovery of Physical Function After Critical Illness In Older Adults
Acronym: RETURN
Status: Not yet recruiting | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Kirby Mayer, Associate Professor, University of Kentucky
Other Study IDs: 106867
Record Dates: First submitted 2025-10-01; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Acute Lung Injury(ALI)
Keywords: sepsis; acute respiratory failure; intensive care unit; Acquired muscle weakness
MeSH Terms: conditions — Sepsis; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and muscle tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RETURN: Survivors of critical illness

SUMMARY:
The proposed study is a prospective, observational study assessing the recovery of muscle and physical function in patients surviving critical illness (n =150) at hospital discharge (baseline) and repeated serially. Patients will be enrolled after life-saving modalities have been weaned near hospital discharge. Patients will participate in testing at baseline, 3-, 6-, 12-, and 24-months after hospital discharge. In a subset of patients (n = 18), muscle biopsies will be performed at baseline and then repeated once at either 12- or 24-months after hospital discharge.

DETAILED DESCRIPTION:
The overarching goal of the proposed study is to determine the trajectories of physical recovery and cellular markers involved with the underlying failure to recover muscle after critical illness, while exploring which characteristics are associated with sustained physical disability. This proposal will examine muscle pathophysiology carefully aligned with physical function outcomes in order to longitudinally assess the recovery, or failed recovery, of muscle function in participants after critical illness:

Aim 1: Determine the long-term trajectory of muscle strength, physical function and ADL recovery in ICU survivors. Patients (n = 150) will participate in a battery of tests to determine muscle and physical function aligned with self-reported measures of ADLs and quality of life at hospital discharge, 3-, 6-, 12-, and 24-months post.

Aim 2: Assess cellular changes in skeletal muscle in ICU survivors contributing to long-term physical dysfunction. In a subgroup of patients enrolled in Aim 1, muscle biopsies will be collected at baseline and long-term follow-up to determine oxidative stress, mitochondrial function, and cellular senescence.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥40 years of age)
* patients who have survived an ICU admission of at least 72 hours
* diagnosis of acute lung injury or sepsis are eligible.

Exclusion Criteria:

* individuals who were not ambulatory prior to ICU admission,
* not expected to survive at least 6 months,
* have a new or pre-existing brain infarct, injury, or neurological condition with deficits preventing participation in physical testing,
* have a pre-existing geriatric syndrome that were confound recovery trajectory

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of acute lung injury or sepsis who have survived an Intensive Care Unit admission for at least 72 hours.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-05-31 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength measured by Chair Rise Test | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Performance on 5x sit to stand test will be the primary outcome measure representing lower extremity muscle strength ; measured as time in seconds to complete 5 repetitive sit-stands.
Functional Capacity | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  The 6-minute walk test (6MWT), which measures the distance a participant can walk in six minutes and serves as an indicator of cardiopulmonary function, will be used as a primary outcome.

SECONDARY OUTCOMES:
Muscle morphology # 1 | Percent change from baseline to 12 months
  Myofiber size
Muscle morphology #2 | Percent change from baseline to 12 months
  Myofiber type
Lower-extremity Muscle Power | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Muscular Power: Power will be assessed using a linear potentiometer (HUMAC-360, CSMi, Stoughton, MA) to record the velocity and peak-velocity of a functional movement using a Shuttle MiniPress (Shuttle Systems, Bellingham, WA) as hamstring/gluteal pressdown. Outcome measure is Watts.
Muscle Size and Quality measured by Ultrasound | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Ultrasound imaging will be performed to acquire images of quadriceps and tibialis anterior to measure muscle cross-sectional area, muscle thickness and echo intensity of muscles.
Activities of Daily Living (ADL) | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Katz ADL will be used to assess ADL. The range of scores are 0 - 6 with a higher score being an better outcome.
Health Reported Quality of Life | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  5 Dimension Euro-Quality of Life (EQ-5D) is a self-report instrument including 5 questions and a visual analog scale (0-100) used to measure subjective quality of life with a higher score being a better outcome.
Fatigue | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  The Functional Assessment of Chronic Illness Therapy (FACIT-fatigue instrument) will be used to measure subjective fatigue and quality of life. All items are summed to create a single score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning and a higher quality of life.
Physical Frailty | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Physical frailty will be quantified using Fried Frailty Phenotype with five criteria (weight loss, weakness, exhaustion, gait speed, and physical activity) and the Clinical Frailty Scale. Scoring is 0-5 with: ≥3/5 criteria met indicates frailty; 1-2/5 indicates pre-or-intermediate frailty; 0/5 indicates non-frail.
Physical Activity | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Patients will wear an Actigraph (Garmin, Vivofit 4) or an Oura ring to measure the number of steps per day. The outcome measure will be average number of steps per day over a seven day period.
Muscle strength of quadriceps | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Strength of quadriceps muscle will be recorded using a hand-held dynamometry, Lafayette Manual Muscle Test System Model-01165 (Lafayette Company, Lafayette, IN). Outcome is measured in kilograms.
Grip Strength | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Hand grip strength will be assessed with a handgrip dynamometry (HGD), Jamar Hydraulic dynamometer (Sammons Preston Rolyan, Bolingbrook, IL, USA). Outcome is measured in kilograms (kgs).
Physical function | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  The Short Physical Performance Battery (SPPB) assesses balance, repeated sit-to-stand performance, and 4-meter gait speed. Each component is scored and converted to an ordinal scale, with the total score ranging from 0 to 12.
Physical function | Baseline and repeated 3-, 6-, 12-, and 24-months after baseline assessment.
  Timed-up and Go Test (TUG), which is a measure of mobility and fall risk requiring patients to stand from a chair and walk short-distance for time in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Kirby P Mayer, DPT, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky 40536, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.